CLINICAL TRIAL: NCT06711692
Title: Natural History and Standards of Care in Duchenne Muscular Dystrophy - the U.K. NorthStar Clinical Network.
Brief Title: The U.K. NorthStar Clinical Network
Acronym: NS
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Muscular Dystrophy UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 242567
Record Dates: First submitted 2024-11-08; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne Muscular Dystrophy; NorthStar Clinical Network; Northstar; Standards of care in DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DMD children and adult: Paediatric and adults with DMD

SUMMARY:
The goal of this natural history study is to capture the natural history of Duchenne Muscular Dystrophy (DMD) in children and adults in the United Kingdom. Children and adults with DMD will be invited to join.

The primary objective of the study is to collect longitudinal data on motor and respiratory function in DMD patients from childhood to adulthood.

The secondary objectives of the study include collection of longitudinal data on other aspects of natural history on DMD, including respiratory, cardiac and endocrine complications, neurodiversity (cognitive impairment, neuro-behavioural disorders such as ADHD and autism), changes to bone density and occurrence of fractures, changes to puberty, incidence of scoliosis, unplanned hospital admissions, and quality of life. The study will also collect information on ethnicity.

Participants will attend an annual or bi-annual neuromuscular clinic, and will have a series of assessments and questionnaires with the study team. These include: key medical data, physiotherapy data, respiratory assessments, Quality of Life questionnaires, and DMD questionnaires. Following assessments and questionnaire completion, data is input into the study's tailor-made National Neuromuscular Database.

DETAILED DESCRIPTION:
This study will make use of the existing NorthStar network to collect a wider range of clinically relevant data from paediatric and adult DMD patients, to describe more completely the natural history of the disease in different domains and across different life stages and disease phases. Data will be collected using assessment techniques and outcome measures appropriate to the major phases of the disease, and which are in some cases not currently part of the standard of care for DMD in the UK. The National Neuromuscular Database will continue to be used to collect and store these data. This study will allow the network to continue to describe the current natural history in DMD prospectively, with more robust subject ascertainment and completeness. This will help meet the current need for contemporary natural history data for the evaluation of new therapies, and further research in DMD.

ELIGIBILITY:
Inclusion Criteria:

* All patients with genetically confirmed diagnosis of Duchenne Muscular Dystrophy in the United Kingdom. Recruitment will also be possible in cases in whom the DMD diagnosis is made after a muscle biopsy even if the dystrophin gene variant is still being investigated.

Exclusion Criteria:

* Involvement in clinical trials is not an exclusion criterion nor having had surgical procedures, as this is an observational research study. The regular clinical data of patients in clinical trials will be acquired as part of the clinical follow up.
* Patients based outside of the United Kingdom.

Max Age: 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: DMD patients of all ages (both paediatric and adult) will be recruited into the study. No age limits or restrictions within the DMD population have been set for this study, as the study aims to capture the natural progression or DMD irrespective of the stage of the disease. All DMD patients in paediatric or adult clinical care will therefore be eligible to participate providing they have consented
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Longitudinal data on motor function in Duchenne Muscular Dystrophy (DMD) patients from the childhood to the adult phases of life | From enrolment to the end of the study, across 18 months
  Measure: NorthStar Ambulatory Assessment (NSAA). a scale from 0 (unable), 1 (completes independently but with modifications), and 2 (completed without compensation). Total score 0 - 34 with a higher score denoting a higher level of function.

SECONDARY OUTCOMES:
Longitudinal data on quality of life in childhood and adult patients. | From enrolment to the end of the study, across 18 months
  Measure: Duchenne Muscular Dystrophy Quality of Life Measure (DMD-QoL). The DMD-QoL has a hierarchical (or 'higher-order') factor structure, with 3 lower-order factors (physical, social, and psychological) and 1 higher-order factor (overall quality of life [QoL], comprised of the 3 lower-order factors). Higher scores represent a more positive QoL (overall or within each subscale).
Longitudinal data on quality of life in childhood and adult patients. | From enrolment to the end of the study, across 18 months
  Measure: The Quality of Life in Genetic Neuromuscular Disease Questionnaire (QoL-gNMD). The QoL-gNMD domain is measured on a T score metric i.e. a normal distribution with a mean of 50 and a standard deviation of 10.
  High values represent good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Francesco Muntoni, FRCPCH FMed Sci, Study Chair — University College, London; Professor Giovanni Baranello, MD, PhD, Study Director — University College, London; Professor Michela Guglieri, MD, Study Director — Newcastle University; Professor Rosaline Quinlivan, MD, Study Director — University College, London
Locations (25):
- United Kingdom (25):
  - Aberdeen, NHS Grampian, Aberdeen
  - Belfast Health and Social Care Trust, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Birmingham Community Healthcare NHS Foundation Trust, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - University Hospitals Bristol and Weston, Bristol
  - Cambridge University Hospitals, Cambridge
  - Cardiff and Vale University Health Board, Cardiff
  - NHS Dundee - Tayside, Dundee
  - NHS Greater Glasgow and Clyde, Glasgow
  - Lancashire Teaching Hospitals NHS Foundation Trust, Lancaster
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Alder Hey Children's Hospital Trust, Liverpool
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Evelina London Children's Hospital, London
  - Manchester University NHS Foundation Trust, Manchester
  - Newcastle Hospitals NHS Foundation Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry
  - Oxford University Hospitals, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Swansea Bay University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised summary-level data can be made available on request for collaborations. The data dictionary is currently publicly available.
Supporting Information: CSR
Time Frame: After the study has closed, a clinical study report, publications etc may be shared with researchers. Summary-level anonymised data can be requested, subject to approval.
Access Criteria: Academic researchers may contact the study central research group to request collaboration, usage of assessments, summary level of data.

REFERENCES:
- See also: Funder programme brief — https://www.musculardystrophyuk.org/research/current-projects/northstar-programme/
- See also: GOSH Project Outline — https://www.gosh.nhs.uk/wards-and-departments/departments/clinical-specialties/dubowitz-neuromuscular-centre-dnc-information-parents-and-visitors/dubowitz-neuromuscular-centre/northstar-project/